CLINICAL TRIAL: NCT05052463
Title: Electrolyte Imbalance Analysis at Icu Admission : Retrospective Study
Brief Title: Electrolyte Imbalance Analysis at Intensive Care Unit Admission : Retrospective Study
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, ESRA OZAYAR, Head of Anesthesiology and Reanimation Department, Kecioren Education and Training Hospital
Other Study IDs: erbil elektrolit
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Electrolyte Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- sodium (hypo-hyper-normonatremia)
  Interventions: Other: electrolyte imbalance analysis
- potassium (hypo-hyper-normokalemia)
  Interventions: Other: electrolyte imbalance analysis
- calcium (hyper-hypo-normocalcemia)
  Interventions: Other: electrolyte imbalance analysis
- magnesium (hyper-hypo-normocalcemia)
  Interventions: Other: electrolyte imbalance analysis
- phosphor (hypo-hyper-normophosphatemia)
  Interventions: Other: electrolyte imbalance analysis

INTERVENTIONS:
Other: electrolyte imbalance analysis — ın this retrospective study we aimed to evaluate the relationship between the ıcu prognosis and the electrolyte imbalance

SUMMARY:
The type and severity of electrolyte imbalance in patients admitted to the intensive care unit were analyzed.It was evaluated whether these results had an effect on mortality, length of hospital stay, APACHE II scores and ventilator days

ELIGIBILITY:
Inclusion Criteria: all of the ıcu patients -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ıcu patients
Sampling Method: Non-Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
The analysis the electrolyte imbalance in ICU and the relationship between the icu prognosis. | 2 years
  Natremia (Hypo: <136 mmol/L, Normo: 136-145 mmol/L, Hyper: >145 mmol/L) Kalemia (Hypo: <3.5 mmol/L, Normo: 3.5-5.5 mmol/L, Hyper: >5.5 mmol/L) Calcemia (Hypo: <8.8 mg/dL, Normo: 8.8-10.6 mg/dL, Hyper: >10.6 mg/dL) Magnesemia (Hypo: <1.9 mg/dL, Normo: 1.9-2.5 mg/dL, Hyper: >2.5 mg/dL) Phosphatemia (Hypo: <2.5 mg/dL, Normo: 2.5-4.5 mg/dL, Hyper: >4.5 mg/dL)
  The number of patients in all types of electrolyte imbalance will be determined. The effect of the type of electrolyte imbalance on mortality, APACHE-II score and length of invasive ventilation and hospital stay will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Kecioren Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No